CLINICAL TRIAL: NCT06955897
Title: Characterizing Perceived Physical Fatigability in Nusinersen-treated Adolescents and Adults: The SMA EFFORT
Brief Title: Characterizing Perceived Physical Fatigability in Nusinersen-treated SMA
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Biogen (Industry)
Responsible Party: Principal Investigator, Jacqueline Montes, Professor of Rehabilitation and Regenerative Medicine, Columbia University
Other Study IDs: AAAV5804
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: spinal muscular atrophy; neuromuscular disease; nusinersen; fatigability; exercise; SMA; fatigue
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases; Motor Activity; Fatigue | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Walkers: Participants with SMA who are able to walk without assistance.
  Interventions: Other: Observational
- Sitters: Participants with SMA who are unable to walk without assistance, but are able to sit independently.
  Interventions: Other: Observational
- Non-sitters: Participants with SMA who are unable to sit without assistance.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
The purpose of this project is to investigate the utility of the SMA EFFORT, an SMA-specific patient-reported outcome measure, to assess perceived physical fatigability that is anchored to intensity and duration of activities. We aim to characterize perceived physical fatigability (PPF) in a diverse cohort of people with SMA (pwSMA) and evaluate the change of PPF before and after nusinersen dosing.

DETAILED DESCRIPTION:
Fatigue and fatigability are symptoms often experienced by people living with spinal muscular atrophy (pwSMA). Nusinersen is shown to extend survival and improve motor function, but fatigue and fatigability persist. Treated patients report changes in their ability to complete repetitive physical activities but a way for measuring this has not been created. While tests completed in the clinic by individuals with SMA highlight that fatigability is an important part of the SMA experience,we do not fully understand how pwSMA experience fatigability with everyday tasks. Anecdotal reports of pwSMA suggest a waning effect in endurance toward the end of their treatment window, however this change has not been measured.The SMA EFFORT is specifically designed for pwSMA and aims to better understand how they feel when completing daily physical activities.

ELIGIBILITY:
Inclusion Criteria:

1. All types of 5qSMA (homozygous deletion or point mutation of the SMN1 gene and any number of SMN2 copies)
2. Receiving a stable dosing regimen of 12mg nusinersen for at least 6 months

Exclusion Criteria:

1. An injury or surgery within the previous 3 months that would impact their ability to perform in-clinic function and/or fatigability assessments
2. Enrolled in an ongoing clinical trial, or extension study, expanded access program, or long-term registry of an investigational or recently approved medication
3. Receiving adjuvant and/or dual therapy (e.g., muscle-targeted, NMJ, or symptomatic treatments)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 12 years and older, with genetic diagnosis of all types of 5qSMA, treated with nusinersen (12mg) for at least 6 months, will be included.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2026-12-07 (Estimated); Study Completion 2027-02-26 (Estimated)

PRIMARY OUTCOMES:
SMA EFFORT | Baseline, 1 week, 1 month
  The SMA EFFORT is a perceived physical fatigability patient-reported outcome measure (PROM) that provides a percent (PPF%) total score to each participant based on their participation over the past 30 days.

SECONDARY OUTCOMES:
Revised Upper Limb Module (RULM) | Baseline
  The RULM is used to assess motor function of the shoulder, mid-level elbow, wrist, and hand.
Hammersmith Functional Motor Scale Expanded (HFMSE) | Baseline
  The HFMSE is a 33-item scale designed to assess gross motor function in sitters and walkers with SMA.
Six-Minute Walk Test (6MWT) | Baseline
  The 6MWT is an objective evaluation of functional exercise capacity which measures the maximum distance a person can walk in six minutes over a 25-meter linear course.
Six-Minute Mastication Test (6MMT) | Baseline
  The 6MMT is a measure of chewing endurance in which the individual is asked to continuously chew on a chewing tube for a period of six minutes.
Endurance Shuttle Box and Block Test (ESSBT) | Baseline
  The ESSBT is a test of upper limb function that has been adapted to assess performance fatigability in SMA.
Endurance Shuttle Nine-Hole Peg Test (ESNHPT) | Baseline
  The ESNHPT is used to assess more distal, fine motor upper extremity performance fatigability.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Montes, Pt, EdD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided